CLINICAL TRIAL: NCT03033615
Title: Prospective Review of CT Imaging Data Comparing Quality of Low-Radiation-Dose Images Post-Processed With Iterative Reconstruction Software vs. Machine Learning (AlgoMedica PixelShine) Software
Brief Title: PixelShine vs. Iterative Reconstruction (IR) Processing of CT Images
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: AlgoMedica, Inc. (Industry)
Collaborators: Cedars-Sinai Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: ALG-002
Record Dates: First submitted 2016-11-05; First posted 2017-01-27 (Estimated); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Cancer, Lung; Cancer Liver; X-rays; Effects
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Chest CT (Active Comparator): Conventional processing vs. PixelShine processing
  Interventions: Device: PixelShine; Device: Conventional processing
- Abdominal CT (Active Comparator): Conventional processing vs. PixelShine processing
  Interventions: Device: PixelShine; Device: Conventional processing

INTERVENTIONS:
Device: PixelShine — Machine learning algorithm
Device: Conventional processing — Iterative reconstruction software

SUMMARY:
This study will compare the quality of CT images acquired with very low-dose radiation and processed with commercially available software vs. PixelShine processed images. It would potentially allow imaging facilities to acquire CT scans using lower doses of radiation without sacrificing clarity of CT images. Acquiring high quality CT images with low-dose radiation has the potential to enhance patient safety and has significant implications in imaging practices.

DETAILED DESCRIPTION:
Patients receiving CT scans as part of their standard treatment will be asked to consent to an additional 5 minutes of imaging using very low-dose radiation prior to the conventional-dose CT scan. The prospective review will be performed in two cohorts: Chest CT scans and abdominal CT scans.

Anonymized images will be processed by conventional CT software and compared to the same images processed with machine-learning-based PixelShine. A board-certified radiologist will assess the noise and visual quality of the imaging data.

Study patients will receive approximately 10% more dose than a standard CT scan by participating in the study. There are no known short-term safety issues associated with this study. The study-related very low dose radiation is at a level far below that used for conventional x-ray imaging. The study has been approved by the Radiation Safety Committee as part of the review process.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years of age or older
* Patients must be able and willing to consent to participate in this project
* Patients will be scheduled for a standard of care CT scan

Exclusion Criteria:

* This study does not investigate either a specific disease or a specific patient population-it only examines and compares images obtained at low radiation exposure post-processed with Algomedica's PixelShine software with conventionally processed images
* All other patients will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-08 (Estimated); Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Visual Image Quality as Assessed by Image Noise Reduction | Through study completion, an average of 1 month
  Comparison of image noise

SECONDARY OUTCOMES:
Image Resolution as Assessed by Size of Detected Lesions | Through study completion, an average of 1 month
  Determine smallest size of detectable objects

IPD SHARING:
Plan to Share IPD: No